CLINICAL TRIAL: NCT06649851
Title: A Phase 2 Randomized Open-Label Pilot Study of Granulocyte Colony Stimulating Factor (G-CSF) to Preserve Brain Structure and Function Following Standard Chemoradiation in Patients With Newly Diagnosed MGMT-Methylated Glioblastoma
Brief Title: G-CSF After Chemo-radiation in Patients With Glioblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jorg Dietrich, M.D., Ph.D., Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-580
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-08

CONDITIONS: MGMT-Methylated Glioblastoma; Glioblastoma (GBM); Newly Diagnosed Glioblastoma Multiforme
Keywords: MGMT-methylated glioblastoma multiforme (GBM); Newly diagnosed MGMT-methylated glioblastoma multiforme (GBM); Glioblastoma; Glioblastoma Multiforme (GBM)
MeSH Terms: conditions — Glioblastoma | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim; Radiotherapy; Temozolomide; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Chemoradiation combined with G-CSF (Experimental): Per standard of care, participants undergo a 6-week chemoradiation (chemo-RT) cycle followed by a 4-week break. During this 4-week break after chemo-RT, participants receive granulocyte colony stimulating factor (G-CSF) once per day for 5 days (Days 7-11).
  After the 4-week break, as a part of standard care, participants may then receive up to 6 additional 4-week cycles of chemotherapy (temozolomide (TMZ)). During these additional TMZ cycles, participants will receive G-CSF once per day for 3 consecutive days (Days 14-16). G-CSF is injected under the skin (subcutaneously injected) by a study staff member, or self-administered (or a caregiver) can be trained by a study staff member to administer it at home.
  The chemo-RT (radiation therapy and chemotherapy (TMZ)) are standard of care in this study.
  Interventions: Drug: Granulocyte Colony Stimulating Factor (G-CSF); Radiation: Radiation Therapy + Temozolomide
- Standard Chemoradiation (Other): Participants receive standard of care chemoradiation (chemo-RT) which includes an initial 6-week chemo-RT cycle followed by a 4-week break, and up to 6 additional 4-week chemotherapy (temozolomide (TMZ)) cycles.
  Interventions: Radiation: Radiation Therapy + Temozolomide

INTERVENTIONS:
Drug: Granulocyte Colony Stimulating Factor (G-CSF) — Subcutaneously injected study drug; standard target dose of 5-7 µg/kg/d.
  Other Names: G-CSF; Filgrastim; Granix; Neupogen; Zarxio
  Arms: Standard Chemoradiation combined with G-CSF
Radiation: Radiation Therapy + Temozolomide — Standard of care chemoradiation is radiation therapy + Temozolomide (TMZ). Chemoradiation (chemo-RT) includes an initial 6-week cycle, followed by a 4-week break, and up to 6 additional cycles of TMZ.
  Other Names: Chemo-RT; chemoradiation

SUMMARY:
This research study involves the study of granulocyte colony stimulating factor (G-CSF) in patients with MGMT-methylated glioblastoma multiforme (GBM) that are undergoing standard chemoradiation. The study aims to evaluate G-CSF's effects on brain health and cognitive function.

The name of the study drugs involved in this study are:

* G-CSF (also called Filgrastim)
* Temozolomide (TMZ), a standard of care chemotherapy drug

DETAILED DESCRIPTION:
This is an open-label, randomized, phase II clinical study of using G-CSF in patients with newly diagnosed, MGMT-methylated, GBM treated with standard of care radiation with concurrent and adjuvant chemotherapy with temozolomide. The investigators are testing whether G-CSF can reduce the negative side effects from radiation and chemotherapy on brain health. The investigators are specifically testing the effects of G-CSF on brain structure, cognitive function, and general brain health, and the safety and tolerability of G-CSF.

Participants will be randomized, stratified by age, in a 1:1 fashion to receive either standard of care chemo-radiation (chemo-RT) in combination with G-CSF, or standard of care chemo-RT without G-CSF. Treatment with G-CSF will be initiated after chemo-RT and be completed after 6 cycles of adjuvant chemotherapy with Temozolomide.

This study involves screening for eligibility, standard of care radiation therapy and chemotherapy, study treatment and study visits, and follow-up visits. Participants will be in the study for up to 24 months, including 6 weeks of standard of care chemo-RT, up to 7 months of G-CSF treatment (depending on the number of additional chemotherapy cycles given as a part of standard care) and up to 7 months of active follow-up visits after study treatment ends followed by 12 months of survival follow-up.

Up to 60 participants will be enrolled in this study.

Granulocyte colony-stimulating factor (G-CSF) is a protein that stimulates bone marrow to produce stem cells and blood cells and release them into the bloodstream. It is known to have anti-inflammatory and neuroprotective properties (slowing or halting the loss of neurons). G-CSF is also called Filgrastim, and brand names include Granix®, Neupogen®, and Zarxio®. In addition to testing the safety and tolerability of G-CSF, the researchers in this study are testing whether or not G-CSF can protect cells in the brain or enhance repair in the brain after chemoradiation and during chemotherapy. The U.S. Food and Drug Administration (FDA) has not approved G-CSF to support brain health and cognitive function. However, G-CSF has been approved for several decades and in patients with any type of cancer who develop neutropenia (low white blood cell counts) following chemotherapy, including in patients with glioblastoma, or in patients following stem cell transplantation with low white cell blood counts.

The U.S. Food and Drug Administration (FDA) has approved temozolomide as a treatment option for GBM. Temozolomide is given as standard of care chemotherapy in this study.

The radiation therapy used in this study is standard of care and approved by the U.S. Food and Drug Administration (FDA) as a treatment option for GBM.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have confirmed newly diagnosed glioblastoma multiforme (GBM), World Health Organization (WHO) grade 4, IDH wildtype, either by histological or molecular criteria.
* Molecular analysis needs to confirm a positive MGMT promoter methylation status using standard institutional testing methods.
* Treatment needs to involve a planned 6-week course of standard of care radiation therapy with concurrent and adjuvant 6 monthly chemotherapy with temozolomide. Patients scheduled to receive an abbreviated radiation course (e.g., 3 weeks in elderly patients) are eligible.
* Age ≥18 years. GBM is considered a biologically distinct disease in children. Children are excluded from this study but will be eligible for future pediatric clinical trials.
* Karnofsky Performance Status (KPS) > 60, see Appendix A
* No prior cranial irradiation.
* No existing diagnosis of clinical dementia or high clinical suspicion for presence of any neurodegenerative disease (e.g., Alzheimer's Disease, Fronto-temporal Dementia (FTD), Parkinson's Disease, Motor Neuron Disease, etc.) prior to diagnosis of GBM.
* Life expectancy of greater than 6 months.
* Must be able to undergo repeated brain Magnetic resonance imaging (MRI) studies with administration of gadolinium (contrast enhanced brain MRI).
* Participants must have adequate organ and bone marrow function (as defined below) to be able to receive standard chemoradiation therapy:

  * leukocytes ≥2,500/mcL
  * absolute neutrophil count≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin≤ institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT)≤3 × institutional ULN creatinine≤ institutional ULN OR
  * glomerular filtration rate (GFR) ≥60 mL/min/1.73 m2 unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73 m2.

For patients with Gilbert's syndrome, total bilirubin can be ≤ 3xULN.

* For participants with evidence of chronic hepatitis B virus (HBV) infection by history, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen (use of granulocyte colony stimulating factor (G-CSF)) are eligible for this trial.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to G-CSF (Filgrastim associated allergic reactions).
* Participants with uncontrolled intercurrent illness that could influence leukocyte counts, such as severe infection requiring intravenous antibiotics, or known HIV (human immunodeficiency virus), since HIV/AIDS is an immunocompromising disease affecting lymphocyte counts (one of the correlative biomarkers in this study)
* Pregnant women are excluded from this study because of the use of cytotoxic chemotherapy (temozolomide) and radiation, given as part of standard of care in this trial, is of teratogenic potential or has abortifacient effects. Because there is a risk for adverse events in nursing infants secondary to treatment of the mother with cytotoxic chemotherapy, breastfeeding should be discontinued if the mother is treated with cytotoxic chemotherapy.
* Participants must be able to undergo repeated neurocognitive testing in English (or Spanish). As cognitive outcome is one of the main secondary endpoints of this study, the lack of normative and comparison data for non-English or non-Spanish-speaking patients would confound this outcome in our small sample size (see Statistical Analysis Plan for more details). Presence of significant aphasia or any other language impairment at time of diagnosis with GBM is considered an exclusion criterion. Any concerns or questions about a subject's ability to participate in neurocognitive testing can be directed to the study investigators for further discussion and clarification.
* Participants with active thromboembolic event (pulmonary embolism or deep venous thrombosis) or prior thromboembolic event within 6 months prior to diagnosis of GBM may need to be excluded because of possible risks of thromboembolism with the use of G-CSF and will require further discussion with the PI prior to enrollment on a case-by-case basis.
* Participants with the following medical conditions are excluded and not eligible based on elevated risk of G-CSF associated toxicity: Sickle cell disease or sickle cell trait, congenital neutropenia, hematological malignancy (leukemia or myelodysplastic syndrome).
* Patients who are dependent on high doses of corticosteroids equivalent to 8mg of daily dexamethasone or more, or who are expected to be unable to taper steroids post-operatively to a dose of 4mg of dexamethasone or less prior to start of chemo-RT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | From Day 0 (start of chemoradiotherapy (chemo-RT)) to end of treatment (EoT) +30 days, up to 35 weeks total.
  Adverse events (AEs) will be assessed using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. AEs will be listed and tabulated by type and study arm. AEs will also be categorized as study-related or not. The rate of AEs in all participants, both within study arms and overall, will be calculated and reported with exact 95% confidence intervals. All subjects who have completed at least 3 weeks of cranial radiation therapy will be include in the safety analyses.
Change in Brain Volume from Baseline | Screening (completed in Day -28 through Day 0) through up to 7 months after end of treatment (up to 62 weeks total).
  The degree of ventricular volume expansion (measured in % change from baseline) will be assessed by Magnetic Resonance Imaging (MRI), and serving as a surrogate marker for global brain volume loss and compared to a randomized control group. The contra-lesional lateral ventricle will be segmented in 3D Slicer or similar program to calculate the ventricular volume at each time point. Descriptive statistics with 95% CI will be provided for all endpoints and normality of data distribution will be assessed. If needed, Wilcoxon Rank-Sum test will be used to compare changes in ventricular volume expansion from baseline to endpoints between the groups and the Sign-rank tests will be used to evaluate within group changes between time points (two-sample or paired T-test will be used respectively if the data distribution warrants a parametric approach).

SECONDARY OUTCOMES:
Change in Neurocognitive Function (NCF) | Screening (completed in Day -28 through Day 0) through up to 7 months after end of treatment (up to 62 weeks total).
  Measured using a battery of standardized psychometric instruments (HVLT; COWA; TMT A; TMT B; Coding; Wechsler Adult Intelligence Scale; HVLT Delayed Recall; HVLT Recognition) at screening, 1 month after end of chemo-RT, and 6- and 12- months after EoT. 7 cognitive scores will be calculated, 3 for the HVLT and one for each of the other tests. Raw scores for each cognitive metric will be converted to Z-scores using published normative data. A composite score will also be calculated by averaging the 7 test scores for each subject at each time point. Changes from baseline are calculated by subtracting baseline from each of the follow-up scores. Percent change will be calculated as change from baseline divided by baseline. The difference between the pre-treatment baseline and follow-up NCF scores will be determined by the reliable change index (RCI).
Change in Quality of Life (QOL) | Screening (completed in Day -28 through Day 0) through up to 7 months after end of treatment (up to 62 weeks total).
  Participant-reported QOL will be measured using the validated Functional Assessment of Cancer Therapy including Brain Tumor module (FACT-Br). Scores (ranging from 0 to 4) for each domain as well as a total QOL score are calculated. FACT-Br subscales will be combined and analyzed for change in each of the FACT-Br indices, as well as the total score and subjective cognitive function scores. Analysis approach will include regression modeling. Changes from baseline will be calculated by subtracting baseline from each of the follow-up scores. Percent change will be calculated as change from baseline divided by baseline.
Change in Mood using Hospital Anxiety and Depression Scale (HADS) | Screening (completed in Day -28 through Day 0) through up to 7 months after end of treatment (up to 62 weeks total).
  Participant-reported mood will be measured using the Hospital Anxiety and Depression Scale (HADS) . Scores on 2 subscales (ranging from 0 to 21) for each domain are calculated. Scores will be analyzed for change. Analysis approach will include regression modeling. Analysis approach will include regression modeling. Changes from baseline will be calculated by subtracting baseline from each of the follow-up scores. Percent change will be calculated as change from baseline divided by baseline.
Overall Survival (OS) | Screening (completed in Day -28 through Day 0) through 24 months after enrollment.
  Defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive. Data will be listed, tabulated, and presented descriptively using Kaplan Meier plots.
Progression-Free Survival (PFS) | Screening (completed in Day -28 through Day 0) through 24 months after enrollment.
  Defined as the time from randomization (or registration) to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation. Calculated using the Kaplan Meier method.
Time to Progression (TTP) | Screening (completed in Day -28 through Day 0) through 24 months after enrollment.
  Defined as the time from randomization (or registration) to progression, or censored at date of last disease evaluation for those without progression reported. Calculated using the Kaplan Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Jorg Dietrich, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [jdietrich1@partners.org]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation